CLINICAL TRIAL: NCT05686746
Title: Uses of Baricetinib 4 mg or 2mg Versus MMF to Maintain Lupus Remission Randomized Controlled Trial: Outcomes Over 2 Years
Brief Title: Use of Baricitenib to Maintain of Remission
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Hassanien, Associate Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: systemic lupus
Record Dates: First submitted 2022-12-25; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Lupus or SLE; Nephritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Nephritis | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: participant and investigator and outcome assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baricetinib 4 mg (Experimental): 4 mg oral tablet daily
  Interventions: Drug: Baricitinib 4 MG
- Baricetinib 2 mg (Experimental): 2 mg oral tablet daily
  Interventions: Drug: Baricitinib 2 MG
- MMF (Active Comparator): MMF 500 mg tablet twice daily
  Interventions: Drug: MMF

INTERVENTIONS:
Drug: Baricitinib 4 MG — 4 mg oral daily
  Arms: Baricetinib 4 mg
Drug: Baricitinib 2 MG — 2 mg oral daily
  Arms: Baricetinib 2 mg
Drug: MMF — 1000 mg oral daily
  Arms: MMF

SUMMARY:
Baricitinib a selective Janus kinase (JAK) inhibitors 1&2 have been recognized as a potential therapeutic option in systemic lupus (SLE), also known Baricitinib, a JAK inhibitor, has demonstrated efficacy and safety in the treatment of dermatitis and arthritis 1 ; however, no JAK inhibitor studies have been conducted in lupus nephritis (LN) maintain remission to date.

DETAILED DESCRIPTION:
Baricitinib a selective Janus kinase (JAK) inhibitors 1&2 have been recognized as a potential therapeutic option in systemic lupus (SLE), also known Baricitinib, a JAK inhibitor, has demonstrated efficacy and safety in the treatment of dermatitis and arthritis 1 ; however, no JAK inhibitor studies have been conducted in lupus nephritis (LN) maintain remission to date. Objectives: To assess the efficacy and safety of Baricitinib in patients (pts) with LN by dose 4mg versus 2 mg versus MMF 1 gm daily dose.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Lupus nephritis Disease
* Must be able to swallow tablets
* lupus nephritis in remission

Exclusion Criteria:

* antiphospholipid syndrome disease
* thrombosis history
* sever anemia, leukopenia or thrombocytopenia
* impaired liver and renal function

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
proteins creatinine ratio | 3 months
  nephritis
proteins creatinine ratio | 6 months
  nephritis
proteins creatinine ratio | 1 year
  nephritis

SECONDARY OUTCOMES:
complement 3 | 3 months
  serum level
complement 3 | 6 months
  serum level
complement 3 | 1 year
  serum level
anti ds DNA | 3 months
  serum level
anti ds DNA | 6 months
  serum level
anti ds DNA | 1 year
  serum level
ANA | 3 months
  serum level
ANA | 6 months
  serum level
ANA | 1 year
  serum level

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hassanien, MD, Principal Investigator — Assiut University
Locations (1):
- Manal Hassanien, Asyut, Yes, Egypt

IPD SHARING:
Plan to Share IPD: No
after finishing study